CLINICAL TRIAL: NCT04963933
Title: Treatment of Ruptured and Unruptured Wide-Neck Aneurysms With Nautilus™ Device Assisted Occlusion (TORNADO)
Brief Title: A Medical Device to Treat Brain Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoStream Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-262
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Cerebral Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with the device (Experimental): Patients treated with the Nautilus will be followed up
  Interventions: Device: Nautilus endovascular device

INTERVENTIONS:
Device: Nautilus endovascular device — Patients will be treated with the Nautilus Endovascular device followed by treatment follow up for up to 6 months

SUMMARY:
An aneurysm is a bulge in a blood vessel caused by a weakness in the blood vessel wall, usually where it branches. As blood passes through the weakened blood vessel, the blood pressure causes a small area to bulge outwards like a balloon. Most brain aneurysms only cause noticeable symptoms if they burst (rupture). This leads to an extremely serious condition known as a subarachnoid hemorrhage, where bleeding caused by the ruptured aneurysm can cause extensive brain damage and symptoms.

The study aims to evaluate the safety and effectiveness of a medical device to treat brain aneurysms.

DETAILED DESCRIPTION:
Patients will be treated with the Nautilus, then will be followed up for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with intracranial aneurysm

Exclusion Criteria:

* Unstable neurological deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events | 3-6 months
  The rate of participants experiencing death or stroke in treated vascular territory measured using the NIH stroke scale within 3- 6 months follow-up
Probable benefit | 3-6 months
  Rate of stable, successful aneurysm occlusion measured using the Raymond Roy Occlusion Classification at 3-6 months follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- St. Ivan Rilski University hospital, Sofia, Bulgaria
- Paula Stradina university hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No